CLINICAL TRIAL: NCT00221832
Title: Molecular Genetic Screening and Identification of Congenital Arrhythmogenic Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. C. Wolpert, I. Department of Medicine-Cardiology, University Hospital Mannheim, . Department of Medicine-Cardiology, University Hospital Mannheim
Other Study IDs: 0261.5
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2003-10

CONDITIONS: Long QT Syndrome; Hypertrophic Cardiomyopathy; Arrhythmogenic Right Ventricular Dysplasia
Keywords: Long QT Syndrome; Hypertrophic cardiomyopathy; arrhythmogenic right ventricular dysplasia; Short QT Syndrome; Brugada Syndrome
MeSH Terms: conditions — Long QT Syndrome; Cardiomyopathy, Hypertrophic; Arrhythmogenic Right Ventricular Dysplasia; Short Qt Syndrome; Brugada Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — no biospecimens are to be retained.
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is the identification of familial congenital arrhythmogenic disorders and their clinical follow-up.

DETAILED DESCRIPTION:
Molecular genetic screening in patients with:

* supraventricular
* ventricular arrhythmia
* syncopes of unknown origin and/or suspicion of an arrhythmogenic origin
* family members of patients with sudden cardiac death and aborted sudden cardiac death

Examination of patients includes routine testing like electrocardiogram (ECG), sequential ECGs, exercise testing, invasive electrophysiological stimulation, cardiac magnetic resonance imaging, intravenous drug challenge for identification/exclusion of eg Brugada syndrome. Examples are patients with Long QT Syndrome, Short QT Syndrome, Brugada Syndrome, familial atrial fibrillation, WPW-syndrome, arrhythmias due to familial hypertrophic cardiomyopathy or arrhythmogenic right ventricular dysplasia. Blood samples are taken for further molecular genetic screening.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of syncope, abnormal ECG and suspicion of an arrhythmogenic disease
* Patients with long QT syndrome
* Patients with short QT syndrome, shortened QT intervals, borderline shortened QT intervals
* Patients with Brugada syndrome
* Patients with hypertrophic cardiomyopathy
* Patients with arrhythmogenic right ventricular dysplasia

Exclusion Criteria:

* Inability to understand study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patient sampling with history of syncope, aborted SCD, familial sudden cardiac death, high suspicion of familial cardiac arrhythmias.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2003-10; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Borggrefe, Prof., MD, Study Director — I. Department of Medicine-Cardiology
Locations (1):
- University Hospital Mannheim, I. Department of Medicine, Mannheim, Germany